CLINICAL TRIAL: NCT00788047
Title: A Phase 1, Randomized, Open-Label, Two-Way Crossover Study To Evaluate The Steady-State Effect Of Dimebon [PF-01913539] On The Single-Dose Pharmacokinetics Of The CYP2D6 Substrate Dextromethorphan In Healthy Subjects
Brief Title: A Phase 1 Study To Evaluate The Effect Of Dimebon On The Pharmacokinetics Of Dextromethorphan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1451022
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Huntington Disease; Alzheimer Disease
MeSH Terms: conditions — Huntington Disease; Alzheimer Disease | interventions — Dextromethorphan; latrepirdine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regimen A (Reference) (Other)
  Interventions: Drug: Dextromethorphan
- Regimen B (Test) (Experimental)
  Interventions: Drug: Dimebon + Dextromethorphan

INTERVENTIONS:
Drug: Dextromethorphan — Dextromethorphan HCl 30 syrup single dose
  Arms: Regimen A (Reference)
Drug: Dimebon + Dextromethorphan — Dimebon 20 mg tablets given three times daily for 14 days plus Dextromethorphan HCl 30 syrup single dose administered on Day 12
  Arms: Regimen B (Test)

SUMMARY:
This drug-drug interaction study is being conducted to evaluate the potential effect of Dimebon on the pharmacokinetics on dextromethorphan, a probe substrate of the cytochrome P450 2D6 (CYP2D6) enzyme, after multiple dose administration to healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects.
* Extensive or ultra-rapid metabolizers of CYP2D6 substrates, predicted by genotype.

Exclusion Criteria:

* Existence of significant medical conditions that would impact study results or pose unacceptable risks to study subjects.
* Pregnant or nursing females or females of childbearing potential who are unwilling or unable to use an acceptable method of contraception.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Dextromethorphan exposure in combination with Dimebon 20 mg TID relative to Dextromethorphan exposure alone | Day 12

SECONDARY OUTCOMES:
Safety and Tolerability (Adverse Events, Vital Signs, Clinical Labs, Electrocardiograms) | Day 15
Dextrorphan (the metabolite of dextromethorphan) exposure | Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451022&StudyName=A%20Phase%201%20Study%20To%20Evaluate%20The%20Effect%20Of%20Dimebon%20On%20The%20Pharmacokinetics%20Of%20Dextromethorphan